CLINICAL TRIAL: NCT04597736
Title: Biological Collection for the Study of the Relationship Between the Biological Profiles Observed and the Clinical Evolutions Within the Same Cluster of Transmission of the Coronavirus SARS-CoV-2
Brief Title: Relationship Between Biological Profiles and Clinical Evolutions Within the Same Cluster COVID-19 (COVIDCOLLECT)
Acronym: COVIDCOLLECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RBPH 2020 HENQUELL; 2020-A02381-38 (Other: ANSM)
Record Dates: First submitted 2020-10-02; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-09

CONDITIONS: Covid19; Contact Case
Keywords: SARS-CoV-2; COVID19; Confirmed case; Biological collection; contact case; cluster
MeSH Terms: conditions — COVID-19 | interventions — Blood Specimen Collection; Defecation; Urination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cohort (Experimental): Biological collection with nasopharyngeal samples, saliva, blood, stool and urine
  Interventions: Biological: Biological collection with nasopharyngeal samples, saliva, blood, stool and urine

INTERVENTIONS:
Biological: Biological collection with nasopharyngeal samples, saliva, blood, stool and urine — Subjects with a COVID-19 infection and their contact cases (identification according to health insurance criteria, see "Améli.fr") will be offered a clinical evaluation and the takin of biological samples, whether they are hospitalized or via the outpatient screening channel.
  For the main objective: during the Day0 visit, the subjects who agreed to participate in the study will have a clinical evaluation according to a standardized questionnaire and a nasopharyngeal swab, saliva, blood, stool and urine.
  For secondary objectives : longitudinal follow-up will be carried out for 21 days, for index cases and contact cases, whether they have a positive or negative RT-PCR test on D0. A final consultation will be carried out at M3. Nasopharyngeal samples, saliva, blood, stool and urine will be taken on D10 and D21. A blood test will be taken at M3 to carry out a COVID-19 serology.

SUMMARY:
The hypothesis is that from a cluster defined by a confirmed positive case of COVID-19 and its contact cases, it is possible to study the different expressions and clinical evolutions of COVID-19 infection and to explore the biological profiles related to the observed clinical history. Certain biological determinants (virological, immunological, microbological or gentic) could indeed be correlated with the clinical presentation and/or be useful for personalized care.

The main objective is to study the relationship between the biological profiles observed and the clinical evolutions within the same cluster of transmission of the coronavirus SARS-CoV-2 (positive COVID-19 cases and contact subjects).

DETAILED DESCRIPTION:
Subjects with a COVID-19 infection and thei contact cases (identification according to health insurance criteria, see "Améli.fr") will be offered a clinical evaluation and the takin of biological samples, whether they are hospitalized or via the outpatient screening channel.

For the main objective: during the D0 visit, the subjects who agreed to participate in the study will have a clinical evaluation according to a standardized questionnaire and a nasopharyngeal swab, saliva, blood, stool and urine.

For secondary objectives : longitudinal follow-up will be carried out for 21 days, for index cases and contact cases, whether they have a positive or negative RT-PCR test on D0. A final consultation will be carried out at M3. Nasopharyngeal samples, saliva, blood, stool and urine will be taken on D10 and D21. A blood test will be taken at M3 to carry out a COVID-19 serology.

ELIGIBILITY:
Inclusion Criteria:

* Child or adult, no age limit
* Able to give informed consent to participate in research
* If a minor participant: consent of the legal representatives
* If confirmed case COVID-19 (symptomatic or asymptomatic): laboratory result confirming infection with SARS-CoV-2 by RT-PCR or by serology
* If contact case: people identified as a risk contact according to the criteria of the "Amélie.fr" health insurance

Exclusion Criteria:

* Subjects under tutorship, curatorship, deprived of liberty, safeguard of justice
* Refusal of the child
* Refusal of participation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Virological profile | Day 0
  Nasopharyngeal SARS-CoV-2 viral load at day 0 by RT-PCR (in log or ΔCT)
Virological profile | Day 10
  Nasopharyngeal SARS-CoV-2 viral load at day 0 by RT-PCR (in log or ΔCT)
Virological profile | Day 21
  Nasopharyngeal SARS-CoV-2 viral load at day 0 by RT-PCR (in log or ΔCT)
Virological profile (serology) | Day 0
  SARS-CoV-2 serology by enzyme-linked immunosorbent assays or magnetic chemiluminescence enzyme immunoassay (IgG and IgM titers)
Virological profile (serology) | Day 10
  SARS-CoV-2 serology by enzyme-linked immunosorbent assays or magnetic chemiluminescence enzyme immunoassay (IgG and IgM titers)
Virological profile (serology) | Day 21
  SARS-CoV-2 serology by enzyme-linked immunosorbent assays or magnetic chemiluminescence enzyme immunoassay (IgG and IgM titers)
Immunological profile with blood level for markers of inflammation (cytokine) | Day 0
  cytokine panel by flow cytometry or enzyme-linked immunosorbent assay in pg/mL
Immunological profile with blood level for markers of inflammation (cytokine) | Day 10
  cytokine panel by flow cytometry or enzyme-linked immunosorbent assay in pg/mL
Immunological profile with blood level for markers of inflammation (cytokine) | Day 21
  cytokine panel by flow cytometry or enzyme-linked immunosorbent assay in pg/mL
Immunological profile with blood level for markers of inflammation | Day 0
  markers on immune cell subpopulation by RT-PCR or flow cytometry in CT value or %
Immunological profile with blood level for markers of inflammation | Day 10
  markers on immune cell subpopulation by RT-PCR or flow cytometry in CT value or %
Immunological profile with blood level for markers of inflammation | Day 21
  markers on immune cell subpopulation by RT-PCR or flow cytometry in CT value or %
Biochemical profile by blood dosage of CRP | Day 0
  CRP in mg/l
Biochemical profile by blood dosage of CRP | Day 10
  CRP in mg/l
Biochemical profile by blood dosage of CRP | Day 21
  CRP in mg/l
Biochemical profile by blood dosage of CRP | Day 90
  CRP in mg/l
Biochemical profile by blood dosage of ASAT/ALAT | Day 0
  ASAT/ALAT in U/L
Biochemical profile by blood dosage of ASAT/ALAT | Day 10
  ASAT/ALAT in U/L
Biochemical profile by blood dosage of ASAT/ALAT | Day 21
  ASAT/ALAT in U/L
Biochemical profile by blood dosage of ASAT/ALAT | Day 90
  ASAT/ALAT in U/L
Biochemical profile by blood dosage of LDH | Day 0
  LDH in U/L
Biochemical profile by blood dosage of LDH | Day 10
  LDH in U/L
Biochemical profile by blood dosage of LDH | Day 21
  LDH in U/L
Biochemical profile by blood dosage of LDH | Day 90
  LDH in U/L
Biochemical profile by blood dosage of Lactate | Day 0
  Lactate in mg/l
Biochemical profile by blood dosage of Lactate | Day 10
  Lactate in mg/l
Biochemical profile by blood dosage of Lactate | Day 21
  Lactate in mg/l
Biochemical profile by blood dosage of Lactate | Day 90
  Lactate in mg/l
Biochemical profile by blood dosage of D-Dimer | Day 0
  D-Dimer in µg/L
Biochemical profile by blood dosage of D-Dimer | Day 10
  D-Dimer in µg/L
Biochemical profile by blood dosage of D-Dimer | Day 21
  D-Dimer in µg/L
Biochemical profile by blood dosage of D-Dimer | Day 90
  D-Dimer in µg/L
Biochemical profile by blood dosage of Troponin | Day 0
  Troponin in µg/L
Biochemical profile by blood dosage of Troponin | Day 10
  Troponin in µg/L
Biochemical profile by blood dosage of Troponin | Day 21
  Troponin in µg/L
Biochemical profile by blood dosage of Troponin | Day 90
  Troponin in µg/L
Biochemical profile by blood dosage of Ferritin | Day 0
  Ferritin in µg/L
Biochemical profile by blood dosage of Ferritin | Day 10
  Ferritin in µg/L
Biochemical profile by blood dosage of Ferritin | Day 21
  Ferritin in µg/L
Biochemical profile by blood dosage of RAGE | Day 0
  RAGE (receptor of advanced end glycation products) by enzyme-linked immunosorbent assays in pg/mg total protein
Biochemical profile by blood dosage of RAGE | Day 10
  RAGE (receptor of advanced end glycation products) by enzyme-linked immunosorbent assays in pg/mg total protein
Biochemical profile by blood dosage of RAGE | Day 21
  RAGE (receptor of advanced end glycation products) by enzyme-linked immunosorbent assays in pg/mg total protein
Biochemical profile by blood dosage of SUPAR | Day 0
  SUPAR (soluble urokinase plasminogen activator receptor) by enzyme-linked immunosorbent assays in pg/mg total protein
Biochemical profile by blood dosage of SUPAR | Day 10
  SUPAR (soluble urokinase plasminogen activator receptor) by enzyme-linked immunosorbent assays in pg/mg total protein
Biochemical profile by blood dosage of SUPAR | Day 21
  SUPAR (soluble urokinase plasminogen activator receptor) by enzyme-linked immunosorbent assays in pg/mg total protein
Haematological profile by blood dosage of leukocytes | Day 0
  leukocytes in Giga/L
Haematological profile by blood dosage of leukocytes | Day 10
  leukocytes in Giga/L
Haematological profile by blood dosage of leukocytes | Day 21
  leukocytes in Giga/L
Haematological profile by blood dosage of leukocytes | Day 90
  leukocytes in Giga/L
Haematological profile by blood dosage of Red blood cells | Day 0
  Red blood cells in Tera/L
Haematological profile by blood dosage of Red blood cells | Day 10
  Red blood cells in Tera/L
Haematological profile by blood dosage of Red blood cells | Day 21
  Red blood cells in Tera/L
Haematological profile by blood dosage of Red blood cells | Day 90
  Red blood cells in Tera/L
Haematological profile by blood dosage of Hemoglobin | Day 0
  Hemoglobin in g/dL
Haematological profile by blood dosage of Hemoglobin | Day 10
  Hemoglobin in g/dL
Haematological profile by blood dosage of Hemoglobin | Day 21
  Hemoglobin in g/dL
Haematological profile by blood dosage of Hemoglobin | Day 90
  Hemoglobin in g/dL
Haematological profile by blood dosage of Hematocrit | Day 0
  Hematocrit in %
Haematological profile by blood dosage of Hematocrit | Day 10
  Hematocrit in %
Haematological profile by blood dosage of Hematocrit | Day 21
  Hematocrit in %
Haematological profile by blood dosage of Hematocrit | Day 90
  Hematocrit in %
Haematological profile by blood dosage of Mean corpuscular volume | Day 0
  Mean corpuscular volume in fL
Haematological profile by blood dosage of Mean corpuscular volume | Day 10
  Mean corpuscular volume in fL
Haematological profile by blood dosage of Mean corpuscular volume | Day 21
  Mean corpuscular volume in fL
Haematological profile by blood dosage of Mean corpuscular volume | Day 90
  Mean corpuscular volume in fL
Haematological profile by blood dosage of Mean corpuscular hemoglobin | Day 0
  Mean corpuscular hemoglobin in pg
Haematological profile by blood dosage of Mean corpuscular hemoglobin | Day 10
  Mean corpuscular hemoglobin in pg
Haematological profile by blood dosage of Mean corpuscular hemoglobin | Day 21
  Mean corpuscular hemoglobin in pg
Haematological profile by blood dosage of Mean corpuscular hemoglobin | Day 90
  Mean corpuscular hemoglobin in pg
Haematological profile by blood dosage of average corpuscular concentration of haemoglobin | Day 0
  Average corpuscular concentration of haemoglobin in g/dL
Haematological profile by blood dosage of average corpuscular concentration of haemoglobin | Day 10
  Average corpuscular concentration of haemoglobin in g/dL
Haematological profile by blood dosage of average corpuscular concentration of haemoglobin | Day 21
  Average corpuscular concentration of haemoglobin in g/dL
Haematological profile by blood dosage of average corpuscular concentration of haemoglobin | Day 90
  Average corpuscular concentration of haemoglobin in g/dL
Haematological profile by blood dosage of polynuclear neutrophil | Day 0
  polynuclear neutrophil in Giga/L
Haematological profile by blood dosage of polynuclear neutrophil | Day 10
  polynuclear neutrophil in Giga/L
Haematological profile by blood dosage of polynuclear neutrophil | Day 21
  polynuclear neutrophil in Giga/L
Haematological profile by blood dosage of polynuclear neutrophil | Day 90
  polynuclear neutrophil in Giga/L
Haematological profile by blood dosage of polynuclear eosinophils | Day 0
  polynuclear eosinophils in Giga/L
Haematological profile by blood dosage of polynuclear eosinophils | Day 10
  polynuclear eosinophils in Giga/L
Haematological profile by blood dosage of polynuclear eosinophils | Day 21
  polynuclear eosinophils in Giga/L
Haematological profile by blood dosage of polynuclear eosinophils | Day 90
  polynuclear eosinophils in Giga/L
Haematological profile by blood dosage of polynuclear basophils | Day 0
  polynuclear basophils in Giga/L
Haematological profile by blood dosage of polynuclear basophils | Day 10
  polynuclear basophils in Giga/L
Haematological profile by blood dosage of polynuclear basophils | Day 21
  polynuclear basophils in Giga/L
Haematological profile by blood dosage of polynuclear basophils | Day 90
  polynuclear basophils in Giga/L
Haematological profile by blood dosage of lymphocytes | Day 0
  lymphocytes in Giga/L
Haematological profile by blood dosage of lymphocytes | Day 10
  lymphocytes in Giga/L
Haematological profile by blood dosage of lymphocytes | Day 21
  lymphocytes in Giga/L
Haematological profile by blood dosage of lymphocytes | Day 90
  lymphocytes in Giga/L
Haematological profile by blood dosage of monocytes | Day 90
  monocytes in Giga/L
Haematological profile by blood dosage of monocytes | Day 0
  monocytes in Giga/L
Haematological profile by blood dosage of monocytes | Day 10
  monocytes in Giga/L
Haematological profile by blood dosage of monocytes | Day 21
  monocytes in Giga/L
Haematological profile by blood dosage of platelets | Day 0
  platelets in Giga/L
Haematological profile by blood dosage of platelets | Day 10
  platelets in Giga/L
Haematological profile by blood dosage of platelets | Day 21
  platelets in Giga/L
Haematological profile by blood dosage of platelets | Day 90
  platelets in Giga/L
Haematological profile by blood dosage of activated partial thromboplastin time | Day 0
  activated partial thromboplastin time in second/witness
Haematological profile by blood dosage of activated partial thromboplastin time | Day 10
  activated partial thromboplastin time in second/witness
Haematological profile by blood dosage of activated partial thromboplastin time | Day 21
  activated partial thromboplastin time in second/witness
Haematological profile by blood dosage of activated partial thromboplastin time | Day 90
  activated partial thromboplastin time in second/witness
Haematological profile by blood dosage of fibrinogen | Day 0
  fibrinogen in g/L
Haematological profile by blood dosage of fibrinogen | Day 10
  fibrinogen in g/L
Haematological profile by blood dosage of fibrinogen | Day 21
  fibrinogen in g/L
Haematological profile by blood dosage of fibrinogen | Day 90
  fibrinogen in g/L
Haematological profile by blood dosage of factor V | Day 0
  factor V in %
Haematological profile by blood dosage of factor V | Day 10
  factor V in %
Haematological profile by blood dosage of factor V | Day 21
  factor V in %
Haematological profile by blood dosage of factor V | Day 90
  factor V in %

SECONDARY OUTCOMES:
SARS-CoV-2 salivary viral load | Day 0
  RT-PCR SARS-CoV-2 on saliva in ΔCT value or log10 copies per mL
SARS-CoV-2 salivary viral load | Day 10
  RT-PCR SARS-CoV-2 on saliva in ΔCT value or log10 copies per mL
SARS-CoV-2 salivary viral load | Day 21
  RT-PCR SARS-CoV-2 on saliva in ΔCT value or log10 copies per mL
Comparison of viral sequences | Day 0
  bioinformatic and statistical analyzes of viral sequences (arbitrary unit and p-values)
Comparison of viral sequences | Day 10
  bioinformatic and statistical analyzes of viral sequences (arbitrary unit and p-values)
Comparison of viral sequences | Day 21
  bioinformatic and statistical analyzes of viral sequences (arbitrary unit and p-values)
microbiota analysis | Day 0
  bioinformatic and statistical analyzes of microbiota (arbitrary unit and p-values)
microbiota analysis | Day 10
  bioinformatic and statistical analyzes of microbiota (arbitrary unit and p-values)
microbiota analysis | Day 21
  bioinformatic and statistical analyzes of microbiota (arbitrary unit and p-values)
environmental and societal factors (EPICE) | Day 0
  EPICE score (Assessment of precariousness and health inequalities in examination centers Health) at day 0 from 0 to 100
environmental and societal factors | Day 0
  eating habits
environmental and societal factors | day 10
  eating habits
environmental and societal factors | day 21
  eating habits
environmental and societal factors | day 90
  eating habits
environmental and societal factors (SF-36) | Day 0
  SF-36 score (quality of life by Gardenal O) from 0 to 100
environmental and societal factors (SF-36) | day 10
  SF-36 score (quality of life by Gardenal O) from 0 to 100
environmental and societal factors (SF-36) | day 21
  SF-36 score (quality of life by Gardenal O) from 0 to 100
environmental and societal factors (SF-36) | day 90
  SF-36 score (quality of life by Gardenal O) from 0 to 100
environmental and societal factors (Physical activity) | Day 0
  Physical activity score (by J. Ricci et L. Gagnon test for adults and ActiFitY test for children) from 0 to 100
environmental and societal factors (Physical activity) | day 10
  Physical activity score (by J. Ricci et L. Gagnon test for adults and ActiFitY test for children) from 0 to 100
environmental and societal factors (Physical activity) | day 21
  Physical activity score (by J. Ricci et L. Gagnon test for adults and ActiFitY test for children) from 0 to 100
environmental and societal factors (Physical activity) | day 90
  Physical activity score (by J. Ricci et L. Gagnon test for adults and ActiFitY test for children) from 0 to 100
body weight | Day 0
  body weight in kg
body weight | day 10
  body weight in kg
body weight | day 21
  body weight in kg
body weight | day 90
  body weight in kg
oxygen saturation | Day 0
  oxygen saturation in %
oxygen saturation | day 10
  oxygen saturation in %
oxygen saturation | day 21
  oxygen saturation in %
oxygen saturation | day 90
  oxygen saturation in %
Respiratory rate | Day 0
  Respiratory rate per minute
Respiratory rate | day 10
  Respiratory rate per minute
Respiratory rate | day 21
  Respiratory rate per minute
Respiratory rate | day 90
  Respiratory rate per minute
cardiac frequency | Day 0
  cardiac frequency per minute
cardiac frequency | day 10
  cardiac frequency per minute
cardiac frequency | day 21
  cardiac frequency per minute
cardiac frequency | day 90
  cardiac frequency per minute
lung damage | Day 0
  Lung damage on auscultation in terms of presence/absence
lung damage | day 10
  Lung damage on auscultation in terms of presence/absence
lung damage | day 21
  Lung damage on auscultation in terms of presence/absence
lung damage | day 90
  Lung damage on auscultation in terms of presence/absence
lung evolution | day 90
  CT san in terms of normal/abnormal (children and pregnant women not concerned)
blood pressure | Day 0
  Dysatolic/systolic blood pressure in mmHg
blood pressure | day 10
  Dysatolic/systolic blood pressure in mmHg
blood pressure | day 21
  Dysatolic/systolic blood pressure in mmHg
blood pressure | day 90
  Dysatolic/systolic blood pressure in mmHg
body temperature | Day 0
  Body temperature in °C
body temperature | day 10
  Body temperature in °C
body temperature | day 21
  Body temperature in °C
body temperature | day 90
  Body temperature in °C
clinical exam (skin) | Day 0
  Skin mottling in terms of presence/absence
clinical exam (skin) | day 10
  Skin mottling in terms of presence/absence
clinical exam (skin) | day 21
  Skin mottling in terms of presence/absence
clinical exam (skin) | day 90
  Skin mottling in terms of presence/absence
clinical exam (polypnea) | Day 0
  polypnea in terms of presence/absence
clinical exam (polypnea) | day 10
  polypnea in terms of presence/absence
clinical exam (polypnea) | day 21
  polypnea in terms of presence/absence
clinical exam (polypnea) | day 90
  polypnea in terms of presence/absence
denutrition | Day 0
  denutrition in terms of presence/absence
denutrition | day 10
  denutrition in terms of presence/absence
denutrition | day 21
  denutrition in terms of presence/absence
denutrition | day 90
  denutrition in terms of presence/absence
Antibiotic treatment | Day 0
  Antibiotic treatment in terms of presence/absence with precision if necessary
Antibiotic treatment | day 10
  Antibiotic treatment in terms of presence/absence with precision if necessary
Antibiotic treatment | day 21
  Antibiotic treatment in terms of presence/absence with precision if necessary
Antibiotic treatment | day 90
  Antibiotic treatment in terms of presence/absence with precision if necessary
Steroidal anti-inflammatory treatment | Day 0
  Steroidal anti-inflammatory treatment in terms of presence/absence with precision if necessary
Steroidal anti-inflammatory treatment | day 10
  Steroidal anti-inflammatory treatment in terms of presence/absence with precision if necessary
Steroidal anti-inflammatory treatment | day 21
  Steroidal anti-inflammatory treatment in terms of presence/absence with precision if necessary
Steroidal anti-inflammatory treatment | day 90
  Steroidal anti-inflammatory treatment in terms of presence/absence with precision if necessary
Anti-diabetic treatment | Day 0
  Anti-diabetic treatment in terms of presence/absence with precision if necessary
Anti-diabetic treatment | day 10
  Anti-diabetic treatment in terms of presence/absence with precision if necessary
Anti-diabetic treatment | day 21
  Anti-diabetic treatment in terms of presence/absence with precision if necessary
Anti-diabetic treatment | day 90
  Anti-diabetic treatment in terms of presence/absence with precision if necessary
Gastric protector treatment | Day 0
  Gastric protector treatment in terms of presence/absence with precision if necessary
Gastric protector treatment | day 10
  Gastric protector treatment in terms of presence/absence with precision if necessary
Gastric protector treatment | day 21
  Gastric protector treatment in terms of presence/absence with precision if necessary
Gastric protector treatment | day 90
  Gastric protector treatment in terms of presence/absence with precision if necessary
chills | Day 0
  chills in terms of presence/absence
chills | day 10
  chills in terms of presence/absence
chills | day 21
  chills in terms of presence/absence
chills | day 90
  chills in terms of presence/absence
Myalgia | Day 0
  Myalgia in terms of presence/absence
Myalgia | day 10
  Myalgia in terms of presence/absence
Myalgia | day 21
  Myalgia in terms of presence/absence
Myalgia | day 90
  Myalgia in terms of presence/absence
Anorexia | Day 0
  Anorexia in terms of presence/absence
Anorexia | day 10
  Anorexia in terms of presence/absence
Anorexia | day 21
  Anorexia in terms of presence/absence
Anorexia | day 90
  Anorexia in terms of presence/absence
Rhinitis | Day 0
  Rhinitis in terms of presence/absence
Rhinitis | day 10
  Rhinitis in terms of presence/absence
Rhinitis | day 21
  Rhinitis in terms of presence/absence
Rhinitis | day 90
  Rhinitis in terms of presence/absence
Confusion | Day 0
  Confusion in terms of presence/absence
Confusion | day 10
  Confusion in terms of presence/absence
Confusion | day 21
  Confusion in terms of presence/absence
Confusion | day 90
  Confusion in terms of presence/absence
Asthenia | Day 0
  Asthenia in terms of presence/absence
Asthenia | day 10
  Asthenia in terms of presence/absence
Asthenia | day 21
  Asthenia in terms of presence/absence
Asthenia | day 90
  Asthenia in terms of presence/absence
Falls at home | Day 0
  Falls at home in terms of presence/absence
Falls at home | day 10
  Falls at home in terms of presence/absence
Falls at home | day 21
  Falls at home in terms of presence/absence
Falls at home | day 90
  Falls at home in terms of presence/absence
Insomnia | Day 0
  Insomnia in terms of presence/absence
Insomnia | day 10
  Insomnia in terms of presence/absence
Insomnia | day 21
  Insomnia in terms of presence/absence
Insomnia | day 90
  Insomnia in terms of presence/absence
Angina | Day 0
  Angina in terms of presence/absence
Angina | day 10
  Angina in terms of presence/absence
Angina | day 21
  Angina in terms of presence/absence
Angina | day 90
  Angina in terms of presence/absence
Ageusia | Day 0
  Ageusia in terms of presence/absence
Ageusia | day 10
  Ageusia in terms of presence/absence
Ageusia | day 21
  Ageusia in terms of presence/absence
Ageusia | day 90
  Ageusia in terms of presence/absence
Respiratory complaints | Day 0
  Respiratory complaints in term of SRIpr score from 0 to 100
Respiratory complaints | day 2
  Respiratory complaints in term of SRIpr score from 0 to 100
Respiratory complaints | day 4
  Respiratory complaints in term of SRIpr score from 0 to 100
Respiratory complaints | day 6
  Respiratory complaints in term of SRIpr score from 0 to 100
Respiratory complaints | day 8
  Respiratory complaints in term of SRIpr score from 0 to 100
Respiratory complaints | day 10
  Respiratory complaints in term of SRIpr score from 0 to 100
Respiratory complaints | day 21
  Respiratory complaints in term of SRIpr score from 0 to 100
Respiratory complaints | day 90
  Respiratory complaints in term of SRIpr score from 0 to 100
transmission rate | Day 0
  Rate of viral transmission determine by bioinformatic and statistical analyzes in %
transmission rate | day 10
  Rate of viral transmission determine by bioinformatic and statistical analyzes in %
transmission rate | day 21
  Rate of viral transmission determine by bioinformatic and statistical analyzes in %
prolonged viral shedding | between day 0 and day 21
  Prolonged viral shedding evaluate by RT-PCR (CT value or log10 copies per mL)

CONTACTS AND LOCATIONS:
Overall Officials: Céclie Henquell, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France